CLINICAL TRIAL: NCT01643239
Title: Effects of Forms of Modified Constraint-induced Therapy on Functional Performance of Upper Extremity in Children With Cerebral Palsy With Asymmetric Motor Impairments: A Follow up Study of Kinematic and Clinical Analyses
Brief Title: Effects of Forms of Modified CIT on Upper Extremity Performance in Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Collaborators: Chang Gung University (Other); National Science and Technology Council, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 94-1052B
Record Dates: First submitted 2012-07-04; First posted 2012-07-18 (Estimated); Last update posted 2013-02-28 (Estimated); Status verified 2013-02

CONDITIONS: Cerebral Palsy
Keywords: Modified constraint-induced therapy; Children with cerebral palsy; Kinematic analysis; Group therapy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (3):
- Hospital-based mCIT with individualized intervention (Experimental): Hospital-based modified constraint-induced therapy(mCIT)
  Interventions: Other: Hospital-based mCIT restraint of the unaffected arm and practice of the affected arm
- Hospital-based mCIT with group therapy (Experimental): Hospital-based modified constraint-induced therapy(mCIT)
  Interventions: Other: Hospital-based mCIT
- Hospital-based TR (Other): Hospital-based traditional rehabilitation (TR)
  Interventions: Other: Hospital-based TR

INTERVENTIONS:
Other: Hospital-based mCIT restraint of the unaffected arm and practice of the affected arm — the mCIT group with individualized intervention
  Other Names: Hospital-based modified constraint-induced therapy(mCIT)
  Arms: Hospital-based mCIT with individualized intervention
Other: Hospital-based mCIT — the mCIT group with individualized intervention
  Other Names: Hospital-based modified constraint-induced therapy(mCIT)
  Arms: Hospital-based mCIT with group therapy
Other: Hospital-based TR — OT or PT or therapist-based training
  Other Names: Hospital-based traditional rehabilitation (TR)
  Arms: Hospital-based TR

SUMMARY:
The purpose of this study will employ clinical assessment tools to examine the effects of modified constraint-induced therapy (mCIT) on the more affected upper extremity of children with cerebral palsy.

DETAILED DESCRIPTION:
The study included threefold: (1) It will employ kinematic analysis, along with clinical assessment tools to examine the effects of mCIT on the more affected upper extremity of children with cerebral palsy with asymmetric motor impairments after treatment immediately and 1 year following. The clinical tools will include Motor Activity Log (MAL), Bruininks-Oseretsky Test of Motor Proficiency (BOTMP),Peabody-Developmental Motor Scales (PDMS-II), and Wee-FIM. (2) This study looked at the intervention impact on bimanual coordination and the less affected upper extremity. (3) It investigated the effects of forms (group vs. individual intervention) on upper extremity performance.

ELIGIBILITY:
Inclusion Criteria:

1. clinical diagnosis of spastic CP
2. age between 4 and 10 years old
3. shoulder flexion of the affected upper limb more than 90 degrees, elbow extension over 160 degrees, wrist extension to 10 degrees at least, and fingers full flexion to 10 degrees at least
4. basic balance ability: sitting on the chair without arm support; feet stay on the floor consistently; performing the affected upper limb movement without losing balance
5. ability to follow simple oral commands
6. no related musculoskeletal surgery of the affected upper limb
7. not have injected the Botox into the affected upper extremity during the past 6 months
8. no visual or auditory disability

Ages: 4 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 1996-08; Primary Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Kinematic assessment | up to six years
  An analysis program coded by LabVIEW (National Instruments, Inc., Austin, TX) language was used to process the kinematic data. The variables of reaction time (sec), normalized movement time (sec/mm), normalized total displacement (unit), joint ranges recruitment (normalized shoulder flexion angle, normalized elbow flexion; degree/mm) angle, and normalized maximum shoulder abduction angle), and maximum shoulder and elbow cross correlation were collected.

SECONDARY OUTCOMES:
Clinical measures at the motor quality and performance include Motor Activity Log (MAL), Bruininks-Oseretsky Test of Motor Proficiency (BOTMP), and Peabody-Developmental Motor Scales (PDMS-II) | up to six years
  The clinical tools used in this study measure the intervention impact on bimanual coordination and unilateral performance of upper extremity.

CONTACTS AND LOCATIONS:
Overall Officials: Ching-yi Wu, ScD, Principal Investigator — Department of Occupational Therapy, Chang Gung Univ.
Locations (1):
- Chang Gung Memorial Hospital, Kwei-shan, Toayuan County, Taiwan